CLINICAL TRIAL: NCT00486200
Title: A Phase II, Dose-Finding Study With ASP2151 in Subjects With Recurrent Episodes of Genital HErpes
Brief Title: A Study With ASP2151 in Subjects With Recurrent Episodes of Genital Herpes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15L-CL-101
Record Dates: First submitted 2007-06-12; First posted 2007-06-14 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Herpes Genitalis
Keywords: ASP2151; Herpes Genitalis; Sexually Transmitted Disease; Herpes Simplex Virus Genital Infection; Treatment Outcome; Genital Herpes
MeSH Terms: conditions — Herpes Genitalis; Sexually Transmitted Diseases | interventions — ASP2151; Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Active Comparator): Oral administration of active comparator
  Interventions: Drug: valacyclovir
- 2 (Placebo Comparator): Oral administration of placebo
  Interventions: Drug: Placebo
- 3 (Experimental): Dosing regimen 1
  Interventions: Drug: ASP2151
- 4 (Experimental): Dosing regimen 2
  Interventions: Drug: ASP2151
- 5 (Experimental): Dosing regimen 3
  Interventions: Drug: ASP2151
- 6 (Experimental): Dosing regimen 4
  Interventions: Drug: ASP2151

INTERVENTIONS:
Drug: ASP2151 — Oral administration.
  Arms: 3; 4; 5; 6
Drug: valacyclovir — Oral administration of active comparator.
  Arms: 1
Drug: Placebo — Oral administration of placebo.
  Arms: 2

SUMMARY:
A study of ASP2151 in subjects with recurrent outbreaks of genital herpes.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a history of genital HSV documented by laboratory testing at screening
* Subject has experienced 4 or more episodes of genital herpes during the past 12 months

Exclusion Criteria:

* Subject is immunocompromised

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 695 (Actual)
Dates: Start 2007-06-21 (Actual); Primary Completion 2008-08-12 (Actual); Study Completion 2008-08-12 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy and safety of ASP2151 with valacyclovir and placebo in the acute treatment of recurrent genital Herpes Simplex Virus Infection | 17 days

SECONDARY OUTCOMES:
Pharmacokinetics in study patients | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma US, Inc.
Locations (24):
- United States (24):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Los Angeles, California
  - Sacramento, California
  - San Diego, California
  - Westlake Village, California
  - Denver, Colorado
  - Boynton Beach, Florida
  - Miami, Florida
  - Atlanta, Georgia
  - Indianapolis, Indiana
  - Madisonville, Kentucky
  - Baltimore, Maryland
  - Billings, Montana
  - Omaha, Nebraska
  - Albuquerque, New Mexico
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Arlington, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - Annandale, Virginia
  - Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tyring S, Wald A, Zadeikis N, Dhadda S, Takenouchi K, Rorig R. ASP2151 for the treatment of genital herpes: a randomized, double-blind, placebo- and valacyclovir-controlled, dose-finding study. J Infect Dis. 2012 Apr 1;205(7):1100-10. doi: 10.1093/infdis/jis019. Epub 2012 Feb 20. PMID 22351940
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/study.aspx?ID=231